CLINICAL TRIAL: NCT06869694
Title: Diagnostic and Predictive Performance of Dual-/ Muti- Energy CT and MRI in the Treatment Response and Survival Prognosis of Gastric Cancer
Brief Title: Energy CT in Imaging and Diagnosis of Gastric Cancer
Acronym: CTIDGC
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Zihao Zhao, The First Affiliated Hospital of Zhengzhou University, The First Affiliated Hospital of Zhengzhou University
Other Study IDs: PC202409
Record Dates: First submitted 2025-03-06; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2024-09

CONDITIONS: Gastric Cancer; CT
Keywords: CT; Gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- GC group: GC patients under ct and mri scan
  Interventions: Device: computerized tomography

INTERVENTIONS:
Device: computerized tomography — mpMRI and Photon-counting Detector CT scan

SUMMARY:
Accurate preoperative prediction of risk stratification, treatment response, and survival prognosis in gastric cancer is important for improving clinical treatment decisions, prolonging patient survival, and improving patient quality of life. The purpose of this study is to investigate the performance of the multi-parametric magnetic resonance imaging (mpMRI) and Dual-/Muti-energy CT and photon-counting Detector CT(PCD-CT) in the diagnosis and management of gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Pathological biopsy confirmed gastric cancer;
2. Surgery: patients undergoing radical gastrectomy. Patients undergoing exploratory abdominal surgery or palliative tumor resection were still included in the study when peritoneal metastasis or adjacent organ invasion was identified intraoperatively and radical surgical resection was not possible.

Exclusion Criteria:

1. Refusal or inability to sign informed consent;
2. CT or MRI images are poor or the focus is small and CT images are not clear;
3. Patients with other tumors complicated with patients with important organ dysfunction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For patients undergoing radical resection, abdominal exploration or palliative tumor resection, CT scanning and dynamic contrast-enhanced magnetic resonance DCE-MRI scanning shall be completed in GSI mode before operation; for patients undergoing neoadjuvant chemotherapy, CT scanning and dynamic contrast-enhanced magnetic resonance DCE-MRI scanning shall be completed in GSI mode before neoadjuvant chemotherapy at least, and if the above scanning mode can still be used during chemotherapy, it is the best choice.
  Signed informed consent form. Patients who were diagnosed with gastric cancer at various medical centers were included in this study
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic and Predictive performance of Dual-/ Muti- energy CT and MRI in the treatment response and survival prognosis of gastric cancer | 3years
  Accuracy for both imaging techniques in the prediction of treatment response of gastric cancer.

SECONDARY OUTCOMES:
The kappa value; One-way analysis of variance; ICC | 1year
  Consistency of the Photon-counting Detector CT and mpMRI in tumor assessment

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, China, China